CLINICAL TRIAL: NCT03992105
Title: Alternative Device to the Accompaniment Called "Place of Respite" in the Resolution of the Psychotic Crises of the People Without a Severe Mental Pathology
Brief Title: Alternative Care to the Accompaniment Called "Place of Respite" in the Resolution of the Psychotic Crises of Homeless People With Severe Mental Pathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-33
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- historical cohort (Other): 150 homeless patients in crisis, identified from an extraction of the database of psychiatric emergencies of the same territory, and matched for age, sex, and main diagnosis.
  Interventions: Other: prospective cohort

INTERVENTIONS:
Other: prospective cohort — topics included openly in the "Respite Site", made up of the first 50 subjects followed prospectively

SUMMARY:
Document the effectiveness of the "Respite Site" program in relation to the current health system. Document in particular the number and type of constraints, lengths of hospitalization and mode of exit, as well as the exit destination of psychotic homeless people.

DETAILED DESCRIPTION:
Between 2012 and 2015, the practice of "stress-related care" related to crisis situations increased by 15%, with about 90,000 people under duress making France one of the European countries where practice most under stress. Being homeless, from a visible ethnic minority, combined with the lack of alternatives in the territory are well-documented risk factors for being hospitalized under duress. A review of the 2015 literature has shown that out-of-hospital crisis sites achieve results equivalent to those of conventional hospitalization in terms of reduced symptomatology and would have better outcomes in terms of increase in remission and recovery times of professional activity and social inclusion, with greater efficiency. In Marseille, an experimental device has shown its capacity to propose an alternative to hospitalization, for this type of population.Running the lessons of this experiment and inspired by the experimentation Parachute, a new device experimental, called "Place of respite", This place proposes a model of resolution of the psychotic crisis where the person decides the type of care that she wish to receive. It is a device that is therefore an alternative to conventional psychiatric care under duress. The investigators formulate the hypothesis that alternative support to the resolution of the crisis by using the skills of people with disorders severe psychiatric conditions in the experimental "Respite site" decreases in the short term the number of hospitalizations and their duration, as well as the experience of the constraint in the course of care of these people, compared to the subjects who did not benefit from this device and could represent a model of crisis management / psychiatric emergency efficient with regard to the current offer.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old Diagnosed with schizophrenia, bipolar I disorder, or schizoaffective disorder according to the DSMIV classification Homeless "ETHOS 1 or 2" (FEANTSA classification) In a crisis situation: psychiatric crisis (PANSS increase of more than 20%), social crisis (significant alteration of social relations) Affiliated to a social protection scheme Accepting to participate in the study An HCAT score greater than or equal to 3

Exclusion Criteria:

Under 18 years old Participant in another study simultaneously in accordance with Article L112112 of the public health code Refusing to participate in the study, or whose legal representative refuses to participate in the study in the case of a person under guardianship or curatorship A score on the HCAT scale (decision-making competence) strictly less than 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Needs Assessement | 36 months
  Scoring the Montreal Assement Need questionnaire